CLINICAL TRIAL: NCT02803229
Title: Treatment of Cannabis Use Disorder Among Adults With Comorbid Attention-Deficit/Hyperactivity Disorder
Acronym: MJ-ADHD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7280; U54DA037842-01 (NIH)
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Cannabis Use Disorder; Attention-deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — SLI381

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): matched Placebo arm
  Interventions: Drug: Matched placebo
- Adderall-XR (Experimental): Adderall-XR (MAS-XR) 80 mg/day maximum maintenance dose
  Interventions: Drug: Adderall-XR

INTERVENTIONS:
Drug: Adderall-XR
  Other Names: Extended-release mixed amphetamine salt
  Arms: Adderall-XR
Drug: Matched placebo — matched placebo provided for placebo arm
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The proposed protocol is a double-blind, placebo-controlled outpatient study of the safety and benefit of Extended-release mixed amphetamine salt (Adderall-XR, MAS-XR) in the treatment of individuals with Cannabis Use Disorder (CUD) and Attention-deficit/Hyperactivity Disorder (ADHD). The investigators plan to enroll 50 and randomize 40 of these patients in the trial. The primary objective of the study is to determine the efficacy of MAS-XR in promoting cannabis abstinence among individuals with CUD and in promoting a decrease of ADHD symptoms.

DETAILED DESCRIPTION:
ADHD is common in substance use disorder patients in general and cannabis use disorder (CUD) in particular, occurring at rates substantially greater than in the general population. A meta-analysis found that approximately 23% of substance abusers seeking treatment have childhood and/or adult ADHD. Moreover, ADHD was overrepresented in adults with CUD compared to other substance use disorder patients seeking treatment. The importance in treating CUD individuals who also have ADHD is underscored by findings demonstrating that individuals with co-occurring ADHD and substance use disorders are a particularly intractable group: they exhibit earlier onset of use, more severe use, a more complicated pattern of remission/relapse, and poorer treatment outcomes relative to those without ADHD. Yet, to date, ADHD individuals with CUD have not been adequately studied. The investigators have found that in their treatment research studies targeting cannabis dependence that a substantial percentage (35%) have screened positive for adult ADHD, rates that are higher than participants in their cocaine use disorder clinical trial and almost 8x greater than rates found in the general population. Thus, this appears to be a sizable cannabis-abusing group warranting much greater clinical attention than they are currently receiving.

The goal is to demonstrate feasibility, tolerability, and estimate effect size for purposes of planning future more definitive trials. Because of the research team's extensive experience in working with stimulant medication in treating ADHD in cocaine-dependent populations, the large effect size of amphetamine in treating adult ADHD, and notable reduction in cocaine use and ADHD symptoms in cocaine-dependent ADHD adults, the investigators will explore the efficacy of Adderall-XR (MAS-XR) for the treatment of cannabis use disorder and ADHD. The study is a 12 week placebo controlled double-blind trial. The maximum maintained dose will be 80 mg of MAS-XR daily.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who meet criteria for cannabis use disorder (CUD) and report that marijuana is their primary drug of abuse
* Individuals must report using marijuana at least 5 days a week over the past 28 days and have a positive urine test for tetrahydrocannabinol (THC) on the day of study entry
* Individuals must meet Diagnostic and Statistical Manual 5th ed. (DSM-5) criteria for adult ADHD
* Individuals who score > 22 on the adult ADHD Investigator Symptom Rating Scale (AISRS)
* Individuals between the ages of 18-65 capable of giving informed consent and capable of complying with study procedures
* Women of child-bearing age will be included if they: a) are not pregnant, b) agree to use an effective method of contraception, c) agree not to become pregnant during the study and d) are not breastfeeding. To confirm this, urine pregnancy tests will be repeated every month after screening. Women will be provided a full explanation of the potential dangers of pregnancy while taking MAS-XR. If a woman becomes pregnant, she will be taken off medication and continue standard treatment. At the end of the study, patients will be offered treatment until an appropriate referral can be made to a community clinic.

Exclusion Criteria:

* Individuals meeting DSM-5 criteria for schizophrenia, schizoaffective illness, psychotic disorder other than transient psychosis due to drug abuse, current major depression, bipolar illness or psychiatric disorders (other than substance abuse) which require psychiatric intervention or would interfere with study participation
* Individuals who are medically unstable based on laboratory tests, electrocardiogram, medical history, physical examination that would make participation hazardous
* Use of synthetic cannabinoids in the past month and meeting CUD diagnosis based on synthetic cannabinoids use alone in the past year
* Individuals with liver enzyme function tests greater than 3 times normal
* Individuals with significant current suicidal risk
* Individuals with systolic blood pressure > 140; diastolic blood pressure >90; pulse >100
* Individuals who are cognitively impaired to impede study participation
* Nursing mothers and pregnant women
* Individuals who are physiologically dependent on any other drugs (excluding nicotine) that would require a medical intervention
* Individuals with known sensitivity/allergy to MAS-XR or amphetamine analogs
* Individuals currently being prescribed psychotropic medication (including sleep medication)
* Individuals with history of seizures
* Individuals who are mandated to treatment
* Individuals with a history of amphetamine use disorders, including amphetamines such as methamphetamine and methylenedioxymethamphetamine (MDMA).
* Individuals with a current cocaine use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, MD, Principal Investigator — New York Psychiatric Institute
Locations (1):
- New York Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study contained a one week placebo lead-in prior to randomization. Three participants were excluded due to being a placebo-responder and two participants were lost to follow-up during this lead-in week.
Groups:
- Adderall-XR: Adderall-XR (MAS-XR) 80 mg/day maximum maintenance dose
  Adderall-XR
Period: Overall Study
Arm/Group | Placebo | Adderall-XR
Started (5 participants were not randomized following the placebo lead-in week.) | 15 | 13
Completed | 11 | 7
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adderall-XR | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (9.5) | 32.4 (11.2) | 32.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 3 | 2 | 5
  White | 8 | 5 | 13
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28
baseline cannabis use [Mean (Standard Deviation); unit: days] — Number of days of self reported cannabis use during 28 days prior to study enrollment.
  days | 26.9 (1.7) | 27.3 (1.1) | 27.1 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Marijuana Abstinence
Description: Number of participants who achieve abstinence from marijuana during the last two weeks of the trial as recorded by the Timeline Followback method and confirmed by urine toxicology.
Time Frame: Change from baseline compared to last 2 weeks of the 12 week study on maintained dose (weeks 10 and 11 for completers) or last 2 weeks of participants' participation during the study for participants who drop out of the study before weeks 10 and 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Adderall-XR
Number analyzed (Participants) | 15 | 13
Participants | 0 | 2

2. Primary Outcome: Reduction in ADHD Symptoms
Description: The primary ADHD outcome measure will be the number of individuals who achieve at least a 30% reduction in symptom severity as measured by the Adult ADHD Interview Rating Scale (AISRS).
Time Frame: Change from baseline compared to last week of trial on maintained dose during the 12 week trial (week 11 for completers) or last week of participants' participation during the 12 week trial for those who drop out of study prior to week 11.
Population: One participant in each arm did not have any follow-up AISRS scores, so they were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Adderall-XR
Number analyzed (Participants) | 14 | 12
Participants | 10 | 10

ADVERSE EVENTS:
Time Frame: 12 weeks of trial or length of participation.
Arm/Group | Placebo | Adderall-XR
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/13
Other Adverse Events (participants affected / at risk) | 5/15 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Adderall-XR (N=13)
Atrial fibrillation (Afib) (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Adderall-XR (N=13)
insomnia (General disorders) | 1 (1) | 3 (3)
anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
chest pain (General disorders) | 0 (0) | 2 (2)
headache (General disorders) | 1 (1) | 1 (1)
nervousness (General disorders) | 1 (1) | 1 (1)
anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
arm numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
backache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dizziness (General disorders) | 0 (0) | 1 (1)
erectile dysfunction (General disorders) | 0 (0) | 1 (1)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
irritability (General disorders) | 0 (0) | 1 (1)
jittery (General disorders) | 0 (0) | 1 (1)
psychomotor agitation (Nervous system disorders) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
tremor (Nervous system disorders) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
weight loss (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT02803229/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT02803229/SAP_001.pdf